CLINICAL TRIAL: NCT05597878
Title: Opioid-Free Pain Control Regimen Following Robotic Radical Prostatectomy: A Randomized Controlled Trial
Brief Title: Opioid-Free Pain Control Regimen Following Robotic Radical Prostatectomy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00091354; WFBCCC 01122 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2022-10-21; First posted 2022-10-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pain Management; Opioid Use; Prostate Cancer
MeSH Terms: conditions — Agnosia; Prostatic Neoplasms | interventions — Oxycodone; Acetaminophen; Ketamine; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Control Cohort (Active Comparator): Participants will receive standard general anesthesia and receive local anesthesia medication (bupivacaine) during surgery per the investigator's surgical protocol. AFTER surgery participants will be administered oxycodone and acetaminophen.
  Interventions: Drug: Oxycodone; Drug: Acetaminophen
- Experimental Non-Opioid Cohort (Active Comparator): Participants will receive standard general anesthesia and receive local anesthesia medication (bupivacaine) during surgery per the investigator's surgical protocol. BEFORE and AFTER surgery participants will be administered Ketamine; DURING surgery Ketorolac and acetaminophen.
  Interventions: Drug: Ketamine; Drug: Ketorolac; Drug: Acetaminophen

INTERVENTIONS:
Drug: Oxycodone — Given after surgery 5 mg every 6 hours as needed for severe pain.
  Arms: Opioid Control Cohort
Drug: Acetaminophen — Given after surgery 1000 mg by mouth 4 times daily (every 6 hours)
  Arms: Opioid Control Cohort
Drug: Ketamine — Given before and during surgery 1.5 mg/kg intravenously
  Arms: Experimental Non-Opioid Cohort
Drug: Ketorolac — Given during surgery 15 mg or 30 mg intravenously 3 times daily (every 8 hours). After surgery 15 mg IV three times daily (every 8 hours).
  Arms: Experimental Non-Opioid Cohort
Drug: Acetaminophen — Given during surgery 1 mg intravenously 4 times daily (every 6 hours). After surgery 1000 mg by mouth four times daily (every 6 hours)
  Arms: Experimental Non-Opioid Cohort

SUMMARY:
The objective of this study is to conduct a randomized clinical trial to evaluate an opioid versus an opioid-free pathway of perioperative use of ketamine, ketorolac, and IV acetaminophen followed by the postoperative use of ketorolac, and oral acetaminophen for pain associated with robotic-assisted radical prostatectomy. Escalation to use of opioid treatment for the opioid-free constituents will be available if needed.

DETAILED DESCRIPTION:
Primary Objective(s): Compare the effectiveness of opioid and opioid-free pathways in treating post-surgical pain following robotic-assisted radical prostatectomy.

Secondary Objective(s)

* To determine the opioid usage in the opioid and non-opioid group from the start of the pain treatment administration until discharge in patients following robotic-assisted radical prostatectomy.
* Determine and analyze preoperative and perioperative measures for opioid and non-opioid groups in patients following robotic-assisted radical prostatectomy.
* Examine and evaluate adverse effects of opioid and opioid-free pathways in patients following robotic-assisted radical prostatectomy using a standardized scale for common post-operative adverse effects including bodily functions.

ELIGIBILITY:
Inclusion Criteria:

* All men ages 40-75 undergoing robot assisted radical prostatectomy (RARP) with or without bilateral lymph node dissection with low, intermediate, or high-risk prostate cancer.
* Patients must have normal organ function as defined below:
* AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
* Creatinine clearance ≥ 30 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Participants with known allergies to any medication involved in the study or its excipients,
* Participants who are incarcerated persons,
* Participants with a chronic narcotic dependence,
* Participants with any prescription for narcotics in the past 30 days,
* Participants who have had only major pelvic or abdominal surgeries as bowel, rectal colon, bladder, liver, gallbladder, kidney, etc. in the past 6 months.
* Patients may not be receiving any other investigational agents.
* Patients with known metastatic disease or brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Scores | Day 0 (prior to surgery); Day 1 (expected hospital discharge) and between days 7-10 (day of postoperative follow up appointment)
  Mean pain scores for opioid and opioid-free groups on Day 0, Day 1, and follow-up appointment between Day 7-10 will be summarized using means and standard deviations. To test that the Day 1 pain levels are not significantly worse in the opioid-free group than in the opioid group, a two sample one sided t-test with a null value of 1.5 for the difference between groups (the non-inferiority margin) will be used. The change in pain from day 0 to days 1, and 7-10 will be compared both within and between groups using t-tests. In addition, a repeated measures linear model, with pain as the outcome and selected demographics and group as covariates, will be used to assess the pain levels and changes in pain across time at all post-operative time points and between groups. Additional preoperative and perioperative covariates will be considered for the model.

SECONDARY OUTCOMES:
Opioid Oral Morphine Milligram Equivalents (OMEQ) | At Day 0 (Prior to surgery) and between Day 7-10 (postoperatively)
  OMEQ will be used to compare opioid use between groups. For continuous measures with skewed distributions, medians and interquartile range will be used as a summary. The comparisons between groups (opioid vs opioid free) will be done using t-tests, Kruskall-Wallis tests, or Chi-squared tests as appropriate.
Demographics of Participants | Day 0 (prior to surgery) to Day 1 (expected hospital discharge)
  Demographics of participants such as age, race will also be used for comparative analysis between groups and will be will be summarized with means and standard deviations or counts and percentages as appropriate.
Preoperative Characteristics of Participants | Day 0 (prior to surgery) to Day 1 (expected hospital discharge)
  Preoperative characteristics such as body mass index, prior abdominal surgeries, cancer risk category, American Society of Anesthesiology (ASA) score, and pre-operative prostate specific antigen (PSA) score will be summarized with means and standard deviations or counts and percentages as appropriate. Perioperative measures such as prostate cancer Grade Group, specimen weight, estimated blood loss, and length of stay (LOS) will also be used for comparative analysis between groups and will be summarized with means and standard deviations or counts and percentages as appropriate.
Opioid-Related Symptom Distress Scale (ORSDS) | Day 0 (prior to surgery); Day 1 (expected hospital discharge) and between days 7-10 (day of postoperative follow up appointment)
  A survey encompassing adverse effects using the Opioid-Related Symptom Distress Scale (ORSDS), will be administered to understand patient's experiences using the medication following robotic-assisted radical prostatectomy on a 4-point scale that evaluates 12 symptoms in 3 symptom categories including frequency, severity, and bother. The ORSDS may be used to calculate a symptom-specific score, which is the average of the 3 symptom distress dimensions and range from 0 to 4. The composite ORSDS score is the mean of all 12 symptom-specific scores. Composite ORSDS scores range from 0 to 4. The ORSDS score will be summarized using means and standard deviations by group.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Hemal, MD, Principal Investigator — Atrium Health Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No